CLINICAL TRIAL: NCT03048955
Title: A 2 and 5 Year Comparative Evaluation of Clinical Outcomes in the Treatment of Moderate Lumbar Spinal Stenosis With the Superion® Indirect Decompression System (IDS) vs. Direct Decompression Surgery for FDA Actual Conditions of Use Study
Brief Title: Assessing Superion Clinical Endpoints vs. Decompression
Acronym: ASCEND
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: FDA and Sponsor closed trial. New post-marketing approval trial in development.
Sponsor: VertiFlex, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-VISS-01
Record Dates: First submitted 2017-01-25; First posted 2017-02-09 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Spinal Stenosis, Lumbar Region With Neurogenic Claudication
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, randomized, controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Indirect Decompression System (Active Comparator): Superion® IDS surgical procedure
  Interventions: Device: Superion® IDS
- Direct decompression Surgery (Active Comparator): Open, direct decompression surgical procedure
  Interventions: Procedure: Direct decompression Surgery

INTERVENTIONS:
Device: Superion® IDS — Device is a non-fusion, spinal column load-sharing device used to stabilize the spine at the implanted leve
  Arms: Indirect Decompression System
Procedure: Direct decompression Surgery — A surgical procedure - the control
  Arms: Direct decompression Surgery

SUMMARY:
PURPOSE: The primary purpose of this study is to demonstrate that the Composite Clinical Success of the study group receiving the Superion® IDS is not inferior to the success rate observed in the study group treated by direct decompression at 60 months follow-up. Secondarily, the trial is intended to establish that Composite Clinical Success of the study group receiving the Superion® IDS at 24 months is not inferior to the success rate observed at 24 months in patients treated with the Superion® IDS in the original IDE trial. Thirdly, the trial is intended to establish that Composite Clinical Success of the population receiving the Superion® IDS in this trial at 24 months is not inferior to the success rate observed at 24 months in patients treated with direct decompression.

DETAILED DESCRIPTION:
STUDY DESIGN:This study is a prospective, multi-center, randomized controlled "Conditions of Use" clinical trial comparing the Superion® IDS to open, direct decompression in the treatment of subjects aged 45 or older suffering from moderate symptoms of neurogenic intermittent claudication secondary to a confirmed diagnosis of moderate LSS at one or two contiguous levels from L1 to L5, i.e. from the L1-L2 level to the L4-L5 level. A maximum of 20 investigative sites in the U.S. will enroll subjects into the trial using a 1:1 randomization assignment. Enrollment will include 358 subjects (152 per arm, plus 18% to account for lost to follow-up). An investigative site is defined as a facility or facilities in the same general geographic location if they are under the control of a local Institutional Review Board (IRB).

After implantation of the Superion® IDS or performance of the direct decompression, each Investigator will be permitted to provide a postoperative care regimen based on the subject's specific need. The regimen may include, but need not be limited to: medications, a corset or brace, acupuncture, traction, physical therapy, chiropractic treatment, use of a TENS unit and massage therapy. The type and amount of the postoperative care will be collected.

At each follow-up visit through 60 months, subjects will be interviewed to determine if they have experienced adverse events (AEs) since the previous follow-up visit. A neurological assessment will be performed for all patients at baseline and all follow-up visits. All subjects will be required to complete ZCQ, ODI, VAS, EQ-5D and the VertiFlex® Patient Satisfaction questionnaires to evaluate disability, function, pain, quality of life and satisfaction at each follow-up visit. Subjects are also required to complete a VAS questionnaire to evaluate pain status at discharge.

The potential impact of spinal injections/nerve blocks use on the ZCQ was evaluated based on review of the medical literature. As these are potentially confounding of the ZCQ outcomes, epidural steroid injections or nerve block procedures at the treated level(s) will be deemed failures. Further, rhizotomy procedures at the treated level(s) will be deemed failures.

With respect to spinal cord stimulators, because the use of a permanent implant would require a surgical procedure, this will be deemed a device failure.

Radiographic evaluations will be performed at discharge, and at each scheduled follow-up visit and prior to any re-operations, in accordance with the Radiographic Evaluation Protocol. The Investigator may also obtain x-rays at unscheduled visits or to assess adverse events, if clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥ 45 years of age.
2. Persistent leg/buttock/groin pain, with or without back pain that is consistently relieved by flexion activities (example: sitting or bending over a shopping cart).
3. Subjects who have been symptomatic and undergoing conservative care treatment for at least 6 months, without relief.
4. Diagnosis of degenerative spinal stenosis of the lumbar spine, defined as the narrowing of the midline sagittal spinal canal (central) and/or narrowing between the facet superior articulating process (SAP), the posterior vertebral margin (lateral access), and the nerve root canal (foraminal).
5. Radiographic confirmation of at least moderate spinal stenosis which narrows the central, lateral, or foraminal spinal canal at one or two contiguous levels from L1-L5. Moderate spinal stenosis is defined as ≤50% reduction in lateral/central foramen.
6. Must present with moderately impaired Physical Function (PF) defined as a score of ≥ 2.0 of the Zurich Claudication Questionnaire (ZCQ).
7. Subjects who are able to give voluntary, written informed consent to participate in this clinical investigation and from whom consent has been obtained.
8. Subjects, who, in the opinion of the Clinical Investigator, are able to understand this clinical investigation, cooperate with the investigational procedures and are willing to return for all the required post-treatment follow-ups.

   * Note: In Criteria #5, all imaging used to confirm LSS should be completed within 4 weeks prior to enrollment. Radiographic confirmation of LSS may include MRI and/or CT.

Exclusion Criteria:

1. Axial back pain only.
2. Fixed motor deficit in lower extremity(ies).
3. Diagnosis of lumbar spinal stenosis which, if the patient were randomized to the Superion arm, would not require any direct neural decompression or surgical intervention other than that required to implant the Superion® device or if randomized to the direct decompression arm, would not require a decompression procedure which would create significant instability requiring spinal fusion, with or without instrumentation.
4. Unremitting pain in any spinal position.
5. Significant peripheral neuropathy or acute denervation secondary to radiculopathy.
6. Lumbar spinal stenosis at more than two levels determined pre-operatively to require surgical intervention.
7. Significant instability of the lumbar spine as defined by ≥ 3mm translation or ≥ 5° angulation through flexion/extension films.
8. Sustained pathologic fractures of the vertebrae or multiple fractures of the vertebrae and/or hips.
9. Spondylolisthesis or degenerative spondylolisthesis greater than grade 1 (on a scale of 1-4).
10. Spondylosis (pars fracture) at the treatment level(s).
11. Degenerative lumbar scoliosis with a Cobb angle of > 10° at treatment level.
12. Osteoporosis, defined as a DEXA bone density measurement T score ≤ -2.5.
13. Morbid obesity, defined as Body Mass Index (BMI) >40kg/m2.
14. Significant peripheral vascular disease (diminished dorsalis pedis or tibial pulses).
15. Prior surgery of the lumbar spine at the treatment level(s).
16. Cauda equina syndrome (defined as neural compression causing neurogenic bowel or bladder dysfunction).
17. Active (systemic, or local in disc or spine) infection at time of surgery.
18. Active systemic disease such as AIDS, HIV, hepatitis, etc.
19. Paget's disease at involved segment or metastasis to the vertebrae, osteomalacia, or other metabolic bone disease.
20. Currently undergoing immunosuppressive therapy or long-term steroid use.
21. Known allergy to titanium or titanium alloys.
22. Tumor in the spine or a malignant tumor except for basal cell carcinoma.
23. Known or suspected history of alcohol and/or drug abuse.
24. Prisoner or transient.
25. Life expectancy less than two years.
26. Any significant psychological disturbance, psychotic or neurotic, that could impair the consent process or ability to complete subject self-report questionnaires.
27. Involved in pending litigation of the spine or worker's compensation related to the back.
28. Enrolled in the treatment phase of another drug or device clinical investigation (currently within past 30 days).
29. Congenital defect of the spine.
30. Pregnant or lactating.
31. Any condition that, in the opinion of the Investigator, would affect the patient's welfare or outcome of the clinical trial.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Composite Endpoint (Primary) | 60 Months
  Subjects in each arm (Superion® IDS and direct decompression) will be evaluated for success at each follow-up interval
Zurich Claudication Questionnaire (ZCQ) | 60 Months
  Clinically significant improvement in outcomes compared to baseline
No re-operations, revisions, removals, or supplemental fixation at the index level(s) | 60 Months
  Review in outcomes compared to baseline
Epidural steroid injections for the treated level(s) | 60 Months
  Review in outcomes compared to baseline

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Coastal Pain Spinal Diagnostics, Carlsbad, California
  - Lake Nona Medical Arts, Celebration, Florida
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - Rothman Institute, Willow Grove, Pennsylvania

IPD SHARING:
Plan to Share IPD: No